CLINICAL TRIAL: NCT07364903
Title: Effectiveness of Implementing Family-Integrated Newborn Care to Improve Outcomes for Preterm and Low-birth-weight Neonates in Resource-limited Settings; Quasi-experimental Design
Brief Title: Effectiveness of Family-Integrated Newborn Care to Improve Outcomes for Preterm and Low-birth-weight Neonates
Acronym: FINC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laerdal Foundation (Other)
Collaborators: Mekelle University (Other); Addis Ababa University (Other)
Responsible Party: Principal Investigator, Znabu Hadush Kahsay, Principal Investigator, University of Stavanger
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LaerdalFoundation
Record Dates: First submitted 2025-12-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Family Involvement/Empowerment; Family-centered Care; Intensive Care Units, Neonatal; Family Integrated Newborn Care
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FINC arm (Experimental): This arm includes the family of the neonates assigned to the experimental group, and they will receive a FINC intervention. The FINC intervention, families of preterm and low-birth weight neonates aged 0-28 days will be trained, educated, and encouraged to get involved in the newborn care targeted to their neonates.
  Interventions: Behavioral: Family Integrated Newborn Care, an intervention to integrate family in the care targeted their preterm and Low-birth weight neonates
- Non-FINC arm (Active Comparator): This arm includes the families of the neonates assigned to the comparator group, who will receive conventional or standard care. No special effort that the routine care will be provided to integrate the family into the care targeted to the preterm and low-birth-weight neonates
  Interventions: Behavioral: Standard medical treatment

INTERVENTIONS:
Behavioral: Family Integrated Newborn Care, an intervention to integrate family in the care targeted their preterm and Low-birth weight neonates — The Family Integrated Newborn Care intervention includes undergoing 1) minor modifications in the NCU space and physical infrastructure conducive to family integration; 2) bedside training for families, and 3) provision of ten audio-visual materials in the local language (Tigrigna) demonstrating family integration in key caring activities targeted to their neonates.
  Other Names: Family-Centered care; Family Involvement
  Arms: FINC arm
Behavioral: Standard medical treatment — The preterm and low-birth weight neonates will receive the conventional care with no special attention to integrate the families in the care targeted to the neonates
  Other Names: Conventional newborn care
  Arms: Non-FINC arm

SUMMARY:
The goal of this quasi-experimental study is to learn if integrating family in newborn care units as a key partner can improve the outcomes of preterm and low-birth-weight neonates. The main question[s] that the study aims to answer:

• Does the implementation of the FINC intervention impact the neonatal outcomes for preterm and low-birth weight neonates in NCUs in resource-limited settings of Tigray, Northern Ethiopia? Researchers will compare the Length of hospital stay among preterm and low-birth-weight neonates admitted to hospitals included in the intervention groups and compared to the neonates admitted to hospitals in the control group.

In the intervention groups, family of preterm and low-birth-weight neonates will be trained, mentored, and integrated into the care targeted to their neonates.

DETAILED DESCRIPTION:
The World Health Organization recommends Family involvement and support in the management of preterm and low birth weight neonates. However, the body of literature on its effectiveness in low-resource settings is scanty. The current study aimed to investigate the effectiveness of implementing Family-Integrated Newborn Care to improve outcomes for preterm and low-birth weight Neonates in resource-limited settings in resource-limited settings of Ethiopia. A quasi-experimental design with non-equivalent comparison groups will be employed among 1020 family-neonate dyads in three hospitals with level-2 Neonatal Care Units. The intervention package will mainly consist of training and education sessions for health care providers and families supplemented by measures to ensure infection prevention in level-2 neonatal care units. The effect size of implementing Family-Integrated Newborn Care on neonatal and parental outcomes will be estimated using General Linear Models (GLM) and compared with the conventional care. Research questions are:

1. Does the implementation of the FINC intervention impact the neonatal outcomes for preterm and low-birth-weight neonates in NCUs in resource-limited settings of Tigray, Northern Ethiopia?
2. Was the uptake of implementation of the FINC intervention for preterm and low-birth-weight neonates acceptable?

ELIGIBILITY:
Inclusion Criteria:

* All neonates aged 0-28 days admitted to level-2 NCUs in the neonatal care unit, including Kangaroo Mother care ward or mothers' side ward, with conditions that require hospital stay at 48 hours; and
* accompanied by at least one parent (preferably a mother) dedicated to spending up to 8 hours per day with the infant

Exclusion Criteria:

* Neonates with major congenital anomalies
* Infants with no family member to accompany the infant, or who do not consent to spend up to 8 hours per day in the NCU
* Families with confirmed physical and/or mental problems limiting their capability to communicate and to engage, or those who leave against medical advice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | The period from the date of admission to the date of discharge is within the first 28 days of neonat's life.
  It refers to the duration a neonate stays in the hospital for care, starting from admission to discharge home

SECONDARY OUTCOMES:
Survival at discharge | Starting from date of admission to the date of discharge within the first 28 days of the neonate's life
  Survival status of the neonate at discharge, specified as alive, dead, or referred for higher-level care, or left against medical advice.
Daily weight gain | Starting from the date of admission up to the date of discharge and assessed in the first 28 days of the neonate's life
  The net weight gain of a neonate each day (in grams/kg/day) in reference to the expected gain for the body mass
Time to initiate breastfeeding after admission | Starting from the date of admission to the date of discharge, within the first 28 days of the neonate's life
  The time the breastfeeding of the neonate is initiated for the first time since admission
Time to initiate skin-to-skin after admission | Starting from the date of admission to the date of discharge, within the first 28 days of the neonate's life
  The first time skin-to-skin is initiated for the neonate, since the date of admission to the Neonatal Intensive Care Unit (NICU)
The number of days on Antibiotics | Starting from the date of admission to the date of discharge, within the first 28 days of the neonate's life
  The total number of days the neonate received antibiotics for being suspected or diagnosed with sepsis
Score for parental stress monitoring scale | Starting from the date of admission to the date of discharge, within the first 28 days of the neonate's life
  A score for the parental stress monitoring scale, which consists of eight items in a five-point Likert scale, with scores ranging from a lower score (1= Not stressful at all) to a higher score (5= Extremely stressful).
Discharge readiness score on the day of the discharge | Starting from the date of admission to the date of discharge, within the first 28 days of the neonate's life
  The score for the discharge readiness scale, consisting of eight items in a five-point Likert scale, to assess parents' readiness at the time of discharge. The score level ranges from a lower score (1= Extremely low confidence) to a higher score (5= Extremely high confidence).

CONTACTS AND LOCATIONS:
Overall Officials: Siren Rettedal, MD, PhD, Study Chair — 1. Faculty of Health Sciences, University of Stavanger, Stavanger, Norway 2. Department of Simulation-based learning, Stavanger University Hospital, Norway; Hege Prof.Ersdal, MD, PhD, Study Director — hege.ersdal@safer.net; Damen Hailemariam, MD, PhD, Study Director — damengoog@gmail.com
Locations (1):
- Mekelle General Hospital, Wukro General Hospital and Adigrat General Hospital, Mek'ele, Tigray, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The study is part of a PhD study. The dataset consists of inpatient data will be shared after the manuscript summarizing the key findings of the trial is published. Hence, the dataset will be made available open for the public in June 2027. In addition, the IPD can be shared up on reasonable request form the contact person of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 2027, one year after the completion of the trial
Access Criteria: The IPD will be available in the data repository for Mekelle University based on the notification to the contact person of the study
URL: https://repository.mu.edu.et/home

REFERENCES:
- [Background] Kahsay ZH, Medhanyie AA, Mariam DH, Ersdal HL, Rettedal S. Feasibility of implementing family-integrated newborn care for hospitalised preterm and low birthweight infants in newborn care units of Ethiopia: a mixed-methods design. BMJ Open. 2025 Jan 21;15(1):e093377. doi: 10.1136/bmjopen-2024-093377. PMID 39842933